CLINICAL TRIAL: NCT01356199
Title: Effet du complément Alimentaire ARTRONAT(R) Sur la réduction de la Gonalgie Chez Des Sujets Arthrosiques
Brief Title: Effect of Artronat on the Quality of Life of Patient With Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lescuyer Laboratory (Industry)
Collaborators: RDVC Produit de Santé. (Unknown); Association Nationale de Prévention Médicale. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2011-A00319-32
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Osteoarthritis
Keywords: Gonalgia; Quality of Life; Dietary supplement; Nutrition
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARTRONAT (Experimental)
  Interventions: Dietary Supplement: ARTRONAT
- PLACEBO (Placebo Comparator)
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: ARTRONAT — Dietary supplement containing Glucosamine, Chondroïtine and manganese. 6 per day for 8 months.
  Arms: ARTRONAT
Dietary Supplement: PLACEBO — PLACEBO. 6 per day for 8 months.
  Arms: PLACEBO

SUMMARY:
The purpose of this study is to determine whether the nutritional supplement ARTRONAT improves the quality of life of patients with osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative disease that greatly impairs the quality of life of patients. A nutritional supplement may help, in association with the normal treatment of osteoarthritis, improving the quality of life of such patients, in reducing pain and/or improving join flexibility.

ELIGIBILITY:
Inclusion Criteria:

* age 40-75 years
* BMI 18.5-30
* osteoarthritis type II or III

Exclusion Criteria:

* osteoarthritis type I or IV
* allergy to one of the component of the supplement
* blood pressure > 14/8
* history of knee surgery

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Reduction of gonalgia | T8 months
  measure with the WOMAC.

SECONDARY OUTCOMES:
Evaluation of the satisfactory relief of symptoms of osteoarthritis at each visit after the beginning of supplementation, assessed by the patients. | T2, T4, T6, T8 months
  Subjective global assessment measured on a 10-cm graduated scale (Visual Analogue Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Cloarec, MD, Study Chair — Association Nationale de Prevention Medicale; Dominique Baron, MD, Principal Investigator — Hospital Center of Lanion
Locations (1):
- Centre Rééducation et Réadaptation Fonctionnelles de Trestel , Centre Hospitalier Pierre-Le-Damany Lannion, Treviou Treguignec, France